CLINICAL TRIAL: NCT04379349
Title: Using Short Message Service as a Means of Clinical Engagement in Early Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, George Foussias, Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 091-2017
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Psychotic Disorders
Keywords: SMS text messaging; Clinical engagement
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active SMS (Experimental): Weekly interactive SMS text messaging check-ins.
  Interventions: Behavioral: SMS text messaging - interactive check-in
- Sham SMS (Sham Comparator): Weekly minimally interactive SMS text messages.
  Interventions: Behavioral: SMS text messaging - inactive control

INTERVENTIONS:
Behavioral: SMS text messaging - interactive check-in — Interactive SMS text message check-ins delivered once weekly to participants.
  Arms: Active SMS
Behavioral: SMS text messaging - inactive control — Minimally interactive SMS text message delivered once weekly to participants.
  Arms: Sham SMS

SUMMARY:
Engagement with clinical services for youth with early psychosis represents a significant challenge, with up to 40% of patients dropping out of treatment in the first year. This has been linked to worse illness outcomes and represents a significant barrier to recovery for these patients. This study aims to evaluate the efficacy of short message service (SMS) as a means of improving clinical engagement in early-episode psychosis populations by bridging contact between appointments with weekly check-ins/reminders. These weekly check-ins during the first year of treatment will serve as an additional opportunity to reach out to patients and give them a chance to do the same with their care teams, with patient responses triggering clinician follow-up if necessary.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 16-29
* a diagnosis of an affective or non-affective psychotic disorder (i.e., Bipolar or Major Depressive Disorders with Psychotic Features, Schizophrenia Spectrum Disorders, Other Specified Psychotic Disorders, Substance Induced Psychosis and Attenuated Psychotic Syndrome)
* eligible for follow-up within the Slaight Family Centre for Youth in Transition early intervention service
* within the first 6 months of treatment

Exclusion Criteria:

* involved in another intervention study
* do not have a personal cell phone number

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Service Engagement Scale (SES) | 9 months
  Clinician-rated treatment engagement and adherence (minimum score = 0, maximum score = 42, higher score indicates worse service engagement)
Appointment Attendance | 9 months
  Percentage of attended clinic appointments

SECONDARY OUTCOMES:
Emergency Department Visits | 9 months
  Number of emergency department visits
Hospitalizations | 9 months
  Number of hospitalizations
Social Functioning Scale (SFS) | 9 months
  Self-report measure of social functioning (minimum score = 0, maximum score = 247, higher score indicates better functioning)
Personal and Social Performance Scale (PSP) | 9 months
  Interview-rated measure of global functioning (minimum score = 1, maximum score = 100, higher score indicates better functioning)
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LESQ-18) | 9 months
  Self-reported measure of subjective quality of life (minimum score = 1, maximum score = 5, higher score indicates better quality of life)
Clinical Global Impression (CGI) | 9 months
  Interview-based global rating of illness severity (minimum score = 1, maximum score = 7, higher score indicates worse illness severity)
Brief Psychiatric Rating Scale (BPRS) | 9 months
  Interview-based measure of the severity of psychiatric symptoms (minimum score = 24, maximum score = 168, higher score indicates higher severity of symptoms)
Scale for the Assessment of Negative Symptoms (SANS) | 9 months
  Interview-based measure of the severity of negative symptoms (minimum score = 0, maximum score = 110, higher score indicates higher severity of symptoms)
Apathy Evaluation Scale (AES) | 9 months
  Interview-rated measure of the severity of motivation deficits (minimum score = 18, maximum score = 72, higher score indicates worse motivation deficits)
Brief Cognitive Assessment Tool for Schizophrenia (B-CATS) | 9 months
  Rater-administered measure of cognitive functioning (scores indicate standardized Z-scores with no pre-defined minimum or maximum score, higher score indicates better cognitive functioning)
Drug Attitude Inventory (DAI-10) | 9 months
  Self-reported measure of medication adherence (minimum score = -10, maximum score = + 10, higher score indicates better adherence)
Scale To Assess Therapeutic Relationships - Patient Version (STAR-P) | 9 months
  Self-reported measure of the clinician-patient therapeutic relationship (minimum score = 0, maximum score = 48, higher score indicates better therapeutic relationship)

CONTACTS AND LOCATIONS:
Overall Officials: George Foussias, MD PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Arcey JN, Zhao H, Wang W, Voineskos AN, Kozloff N, Kidd SA, Foussias G. An SMS text messaging intervention to improve clinical engagement in early psychosis: A pilot randomized-controlled trial. Schizophr Res. 2024 Feb;264:416-423. doi: 10.1016/j.schres.2024.01.012. Epub 2024 Jan 18. PMID 38241785